CLINICAL TRIAL: NCT03496961
Title: Shanghai University of Traditional Chinese Medicine
Brief Title: Yan Nian Jiu Zhuan Fa Improve Chronic Fatigue Syndromes
Acronym: YNJZFCFS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Collaborators: Shanghai Yueyang Integrated Medicine Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 81774443
Record Dates: First submitted 2018-03-19; First posted 2018-04-12 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Chronic Fatigue Syndromes
Keywords: Yan Nian Jiu Zhuan Fa
MeSH Terms: conditions — Fatigue Syndrome, Chronic

STUDY DESIGN:
Intervention Model Description: Clinically evaluated, medically unexplained fatigue of at least 6 months duration:
  Of new onset. Not a result of ongoing exertion. Not substantially alleviated rest and associated with a substantial reduction in previous levels of activity
Who Masked: Participant, Outcomes Assessor
Masking Description: This will use simple randomization ways. Sofware20.0 will used to generate a random unique number for each integral number from 1 to 90 and divide the 90 numbers (1 to 90) into three groups with a ratio of 1:1:1 based on the random numbers group. The number grouping is unknown. This will be a double blind trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Yan Nian Jiu Zhuan Fa (Experimental): The kneading process will be done under the therapist guidance for 30 minutes with an average pressure of 5 Newton each time for 3 times every day.
  Interventions: Behavioral: Yan Nian Jiu Zhuan Fa
- cognitive psychology education (Placebo Comparator): Psychological counseling and behavioral cognition education are conducted once a week and the rest 6 times online or by phone.
  Interventions: Behavioral: Yan Nian Jiu Zhuan Fa
- blank control (No Intervention): this group will have no therapeutic exercises or cognitive education when other two groups receive therapy.

INTERVENTIONS:
Behavioral: Yan Nian Jiu Zhuan Fa — Yan Nian Jiu Zhuan Fa are the kneading methods while cognitive behavior education is the psychological education
  Other Names: cognitive behavior education
  Arms: Yan Nian Jiu Zhuan Fa; cognitive psychology education

SUMMARY:
This study is to disclose the mechanism of characteristic Tao yin exercises regulate Chronic Fatigue Syndromes based on Brain-Gut Axis.Explore the clinical manifestation of Chronic Fatigue Syndromes, changes of neurotransmitter and central brain function. Then provide some new methods of treating Chronic Fatigue Syndromes.

DETAILED DESCRIPTION:
This research will be conducted in Shanghai University of Traditional Chinese Medicine.Then the clinical efficacy of Yan Nian Jiu Zhuan Fa on Chronic Fatigue Syndrome will be observed by examining gastrointestinal function, affecting the content of substances in plasma and analysing the central nerve response mechanism.

ELIGIBILITY:
Inclusion criteria:

The occurrence of four or more of the following symptoms:

* Subjective memory impairment
* Tender lymph nodes
* Muscle pain
* Joint pain
* Headache
* Unrefreshing sleep
* Post-exertion malaise lasting for more than 24 hours

Exclusion criteria:

* Active, unresolved, or suspected medical disease
* Psychotic, melancholic or bipolar depression (but not uncomplicated major depression)
* Psychotic disorders
* Dementia
* Anorexia or bulimia nervosa
* Alcohol or other substance misuse
* Severe obesity.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 135 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Multidimensional Fatigue Inventory (MFI-20) | 6 months
  A self-report instrument consisting of 20-item devised to measure fatigue, covering the dimensions of General Fatigue, Physical Fatigue, Mental Fatigue, Reduced Motivation and Reduced Activity. This instrument takes about 5 to 10 minutes to complete. The instrument's psychometric properties were tested and determined to have good internal consistency and construct validity in samples with Chronic Fatigue Syndrome (CFS).

SECONDARY OUTCOMES:
Short Form 36-item Health Survey (SF-36) | 6 months
  The SF-36 is an internationally well-validated measure of Health-related quality of life that has a broad scope of questions validated across different chronic diseases and comorbidities.
Brain functional connectivity | 6 months
  Functional connectivity density (FCD) is a newly developed data-driven method to measure the number of functional connections of each voxel, possibly providing new insight into the neural correlates of fluid reasoning.Functional magnetic resonance imaging (fMRI) is a novel method for studying the changes of brain functional connectivity.
Bristol Stool Scale | 6 months
  The Bristol stool scale is a diagnostic medical tool designed to classify the form of human feces into seven categories. It is used in both clinical and experimental fields. The seven types of stool are:
  Scale 1: Separate hard lumps, like nuts (hard to pass), also known as goat feces or sausage-shaped, but lumpy.
  Scale 2: Like a sausage but with cracks on its surface or like a sausage or snake, smooth and soft.
  Scale 3: Soft blobs with clear cut edges (passed easily). Scale 4: Fluffy pieces with ragged edges, a mushy stool even watery, no solid pieces, entirely liquid.
  Scale 1 indicate constipation, Scale 2 being the ideal stools as they are easy to defecate while not containing excess liquid, Scale 3 tending towards diarrhea, and Scale 4 indicate diarrhea.
Pittsburgh Sleep Quality Index | 6 months
  A self-report questionnaire that assesses sleep quality over a 1-month time interval. The measure consists of 19 individual items, creating 7 components that produce one global score, and takes 5-10 minutes to complete. Developed by researchers at the University of Pittsburgh, the PSQI is intended to be a standardized sleep questionnaire for clinicians and researchers to use with ease and is used for multiple populations. The questionnaire has been used in many settings, including research and clinical activities, and has been used in the diagnosis of sleep disorders. Clinical studies have found the PSQI to be reliable and valid in the assessment of sleep problems to some degree, but more so with self-reported sleep problems and depression-related symptoms than actigraphic measures.
Neuropeptide Y | 6 months
  Neuropeptide Y (NPY) is a 36 amino-acid neuropeptide that is involved in various physiological and homeostatic processes in both the central and peripheral nervous systems. NPY has been identified as the most abundant peptide present in the mammalian central nervous system, which consists of the brain and spinal cord. It is secreted alongside other neurotransmitters such as glutamate.
Substance P | 6 months
  Substance P is a bioactive 11-amino acid peptide (Arg-Pro-Lys-Pro-Gln-Gln-Phe-Phe-Gly-Leu-Met-amide) first isolated in 1931 from brain and intestine. The peptide is involved in many physiological processes including pain modulation, smooth muscle contraction, blood pressure control, kidney function and water homeostasis.Substance P is widely distributed in numerous tissues and body fluids including the central and peripheral nervous system, gastrointestinal tract, respiratory tract, visual system and circulatory system.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai University of Traditional Chinese Medicine, Shanghai, China

REFERENCES:
- [Result] Bakken IJ, Tveito K, Gunnes N, Ghaderi S, Stoltenberg C, Trogstad L, Haberg SE, Magnus P. Two age peaks in the incidence of chronic fatigue syndrome/myalgic encephalomyelitis: a population-based registry study from Norway 2008-2012. BMC Med. 2014 Oct 1;12:167. doi: 10.1186/s12916-014-0167-5. PMID 25274261
- [Result] Capelli E, Lorusso L, Ghitti M, Venturini L, Cusa C, Ricevuti G. Chronic fatigue syndrome: Features of a population of patients from northern Italy. Int J Immunopathol Pharmacol. 2015 Mar;28(1):53-9. doi: 10.1177/0394632015572074. PMID 25816406
- [Result] May M, Emond A, Crawley E. Phenotypes of chronic fatigue syndrome in children and young people. Arch Dis Child. 2010 Apr;95(4):245-9. doi: 10.1136/adc.2009.158162. Epub 2009 Oct 19. PMID 19843509
- [Result] Porter N, Lerch A, Jason LA, Sorenson M, Fletcher MA, Herrington J. A Comparison of Immune Functionality in Viral versus Non-Viral CFS Subtypes. J Behav Neurosci Res. 2010 Jun 1;8(2):1-8. PMID 24634898
- [Result] Exley C, Swarbrick L, Gherardi RK, Authier FJ. A role for the body burden of aluminium in vaccine-associated macrophagic myofasciitis and chronic fatigue syndrome. Med Hypotheses. 2009 Feb;72(2):135-9. doi: 10.1016/j.mehy.2008.09.040. Epub 2008 Nov 11. PMID 19004564
- [Result] Pardini M, Guida S, Primavera A, Krueger F, Cocito L, Gialloreti LE. Amisulpride vs. fluoxetine treatment of chronic fatigue syndrome: a pilot study. Eur Neuropsychopharmacol. 2011 Mar;21(3):282-6. doi: 10.1016/j.euroneuro.2010.10.008. Epub 2010 Nov 26. PMID 21112746
- [Result] Lloyd S, Chalder T, Rimes KA. Family-focused cognitive behaviour therapy versus psycho-education for adolescents with chronic fatigue syndrome: long-term follow-up of an RCT. Behav Res Ther. 2012 Nov;50(11):719-25. doi: 10.1016/j.brat.2012.08.005. Epub 2012 Aug 31. PMID 22985998
- [Derived] Xie F, Guan C, Gu Y, You Y, Yao F. Effects of the Prolong Life With Nine Turn Method (Yan Nian Jiu Zhuan) Qigong on Brain Functional Changes in Patients With Chronic Fatigue Syndrome in Terms of Fatigue and Quality of Life. Front Neurol. 2022 Jul 13;13:866424. doi: 10.3389/fneur.2022.866424. eCollection 2022. PMID 35911899
- [Derived] Xie F, You Y, Guan C, Xu J, Yao F. The Qigong of Prolong Life With Nine Turn Method Relieve Fatigue, Sleep, Anxiety and Depression in Patients With Chronic Fatigue Syndrome: A Randomized Controlled Clinical Study. Front Med (Lausanne). 2022 Jun 30;9:828414. doi: 10.3389/fmed.2022.828414. eCollection 2022. PMID 35847786
- [Derived] Xie F, Guan C, Cheng Z, Yao F, You Y. Effects of the prolong life with nine turn method (Yan Nian Jiu Zhuan) Qigong on patients with chronic fatigue syndrome: study protocol for a randomized controlled trial. Ann Palliat Med. 2020 Sep;9(5):3571-3583. doi: 10.21037/apm-19-461. Epub 2020 Aug 4. PMID 32787361